CLINICAL TRIAL: NCT02894957
Title: Varenicline for "Gradual" vs. "Abrupt" Smoking Cessation in Low-motivated COPD Smokers: A Randomized Pilot Study
Brief Title: Varenicline for "Gradual" vs. "Abrupt" Smoking Cessation in Low-motivated COPD Smokers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0231-15-SZMC
Record Dates: First submitted 2016-01-31; First posted 2016-09-09 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradual smoking cessation (Experimental): Gradual cessation Patients randomized to the "gradual" cessation group will receive varenicline (0,5 mg once daily for 3 days, 0,5 mg twice daily for 4 days, and 1,0 mg bid thereafter) as an aid for smoking reduction. This pre-treatment phase will last 6 weeks at the end of which all participants must stop smoking altogether. After quitting, they will continue to receive varenicline 1,0 mg bid for a further 12 weeks.
  Smoking reduction: Participants will be recommended to reduce their smoking by 25% in the first two weeks, 50% in weeks 3-4, and 75% in weeks 5-6; however, this will be given only as an indication and every subject will be allowed to chose his/her own goal and rate of progress.
  Interventions: Drug: Varenicline
- Abrupt smoking cessation (Active Comparator): Patients in this group will be asked to smoke as usual for 6 weeks after enrolment then stop altogether. However, those feeling ready will be allowed to quit as of week 4. Thereafter, they will receive the standard 12-week varenicline treatment, starting with a 1 week titration period as described above.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — : Patients will be randomized either to receive varenicline (uptitrated to 1 mg twice daily) for smoking reduction or smoke as usual for 4-6 weeks before quitting. After quit-day, the two groups will receive standard 12-week varenicline treatment. Non-treatment follow-up will continue to 6 months.
  Other Names: champix

SUMMARY:
Rationale: No studies have examined the effect of varenicline for "gradual" smoking cessation in COPD smokers currently not interested in quitting.

Objective: To compare the efficiency of varenicline-assisted "gradual" vs. "abrupt" smoking cessation in low-motivated COPD smokers

Setting: Pulmonary outpatient clinic

Design: Open, randomized pilot smoking cessation trial

Participants: COPD smokers with low motivation to quit. Such low motivation will be defined as a score of ≤ 3 points observed in a 10 cm visual analog scale (0=non motivated; 10=highly motivated).

Interventions/procedures: Patients will be randomized either to receive varenicline (uptitrated to 1 mg twice daily) for smoking reduction or smoke as usual for 4-6 weeks before quitting. After quit-day, the two groups will receive standard 12-week varenicline treatment. Non-treatment follow-up will continue to 6 months.

Measurements: The main outcome measure is carbon monoxide-verified complete abstinence rate (CAR) 6 months after quit-day. Other measures are: CAR at 3 months; point prevalence at 3 and 6 months; change in motivation; cigarettes/day; differential dropout rate; decline in pulmonary function; COPD symptoms, episodes of exacerbation and medication; and adverse events.

Sample size: One hundred twenty-one subjects per group will be necessary to detect CAR differences between the two groups of 15% at 6 months.

Potential study limitations: The main potential limitation is the lack of 1-yr follow-up.

Relevance: This study may provide useful preliminary information on the safety and efficiency of varenicline for "gradual" smoking cessation in low-motivated COPD smokers and it may assist in the preparation of a larger, more comprehensive trial.

DETAILED DESCRIPTION:
RATIONALE

Chronic obstructive lung disease (COPD) is an inflammatory disease characterized by progressive airflow limitation that is not fully reversible by the use bronchodilators .Cigarette smoking is the single most common cause of COPD . It is estimated that 15-20% of smokers will develop COPD over their lifetime, but higher figures have been reported for older smokers. Incidentally, previous studies showed that up to 20% of "healthy" smokers participating in cessation trials might have airway obstruction, most of whom are unaware of this diagnosis . There is no single explanation for the fact that only a fraction of smokers develop COPD. Bronchodilator treatment improves symptoms and quality of life of COPD patients, and new drugs are available for this purpose. Notwithstanding, smoking cessation remains the only therapeutic intervention likely to slow down the progression of the disease by preventing further decline of maximal expiratory flows . Thus, smoking cessation is paramount in the treatment of patients with COPD.

Although they know smoking is the cause of their disease, many patients with COPD continue to smoke. Smoking prevalence rates up to 80 % have been documented in patients with mild to moderate disease and up to 50% in those with severe disease . Notwithstanding, for various reasons COPD patients are more resistant to smoking cessation than "healthy" smokers; these include higher pack-year history and stronger nicotine dependence . In addition, COPD smokers are less motivated to quit and often suffer from depression, a known cause of failure in quit attempts . These observations call for new cessation strategies likely to prompt COPD smokers to attempt to quit smoking.

The standard way to stop smoking is to quit abruptly on a designated quit-day. However, for COPD patients, this can be very hard to achieve since, for them, smoking is not only a source of pleasure but also a longstanding habit, a second nature . An alternative strategy is the so-called "reduce-to-quit" or "gradual" cessation method. Although it also has a quit-day, the key difference is that smokers reduce the number of cigarettes/day over several days or weeks prior to quitting. To help smokers achieve and maintain reduction, pharmacotherapy is usually offered and, in many countries, nicotine replacement therapy (NRT) is licensed for this purpose.

Surprisingly enough, no studies have been published on the efficiency of varenicline as an aid for pre-quitting smoking reduction. Indeed, varenicline was found superior to any single type of NRT (and bupropion) as an aid for smoking cessation in adult smokers. . Second, it was found to be more efficient than placebo and NRT for "abrupt" cessation in COPD smokers motivated to quit ]. Finally, varenicline was found to decrease pre-quit enjoyment in general smokers and increase motivation to quit among healthy smokers who are not willing to make a serious attempt to quit smoking .

RESEARCH QUESTION/OBJECTIVE

With the above considerations in mind, the investigators set out to examine the efficiency of varenicline-assisted "gradual" vs. "abrupt" cessation in COPD smokers with low motivation to quit. The investigators hypothesized that, if these patients received the standard 12-week varenicline treatment, "gradual" cessation would produce higher quit rates at 6 months than "abrupt" cessation if varenicline was used to assist pre-treatment reduction. A secondary hypothesis is that varenicline-assisted pre-quitting smoking reduction would increase motivation to quit compared with usual smoking before quitting.

STUDY DESIGN OVERVIEW

When planning this study, the investigators first idea was to carry out a three-arm, double-blind, randomized trial. However, the lack of basic information for reliable sample size calculation and uncertainties about participation rates guided them towards a preliminary, open, randomized pilot study of COPD smokers with low motivation to quit. The patients will be recruited among those attending the outpatient clinic of Pulmonary Institute of the Share Zedek Medical Center, in Jerusalem. Participants will be randomly assigned to receive varenicline for smoking reduction or smoke as usual before quitting. Thereafter the two groups will receive standard varenicline treatment with follow-up extending to 6 months.

PARTICIPANTS

Participants will be heavy smokers (≥15 pack years) of both sexes, aged ≥35 yrs who received a diagnosis of COPD (FEV1/FVC <70% and FEV1 <80% predicted) with low motivation to quit smoking.

Randomization procedure

Eligible participants will be computer-randomized either to the "gradual" or "abrupt" cessation groups at baseline visit.

Blinding

The study is open so both the participants and the medical team will be aware of treatment.

INTERVENTION AND PROCEDURES

Gradual cessation Patients randomized to the "gradual" cessation group will receive varenicline (0,5 mg once daily for 3 days, 0,5 mg twice daily for 4 days, and 1,0 mg bid thereafter) as an aid for smoking reduction. This pre-treatment phase will last 6 weeks at the end of which all participants must stop smoking altogether. However, patients will be allowed to quit already as of week 4 if they feel ready to do so. After quitting,participants will continue to receive varenicline 1,0 mg bid for a further 12 weeks.

Smoking reduction: Participants will be recommended to reduce their smoking by 25% in the first two weeks, 50% in weeks 3-4, and 75% in weeks 5-6; however, this will be given only as an indication and every subject will be allowed to chose his/her own goal and rate of progress. To achieve reduction each participant will be offered three structured ways: a) Scheduled reduction (SR), that is gradually increasing the time between cigarettes (the inter-cigarette interval); b) Hierarchical reduction - easiest first, that is rating cigarettes in terms of how difficult it would be to give up then eliminate each in turn, starting with the easiest one; and c) Hierarchical reduction - hardest first: this is similar to the previous one but the subject must start by the hardest to give up cigarette first.

Abrupt cessation

Patients in this group will be asked to smoke as usual for 6 weeks after enrolment then stop altogether. However, those feeling ready will be allowed to quit as of week 4. Thereafter, participants will receive the standard 12-week varenicline treatment, starting with a 1 week titration period as described above.

Visits and Follow-up

Ten visits will be scheduled: at study entry and at weeks 2, 4, 6, 8, 10, 14, 18, 24 and 30.

Support

Only minimal levels of advice and support will be given. However, all subjects will receive individualized verbal instructions regarding the general conduct of the study and the proper use of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥35 years
* Currently smoking 10 cigarettes per day or more
* Having smoked 15 py or more
* Presenting a CO level in expired air ≥ 10 ppm
* With low motivation to quit as defined below.
* Willing to sign a statement of informed consent
* Willing to sign a written commitment to quit at a target quit date
* Women of child bearing potential should agree to use acceptable contraception methods.

Exclusion Criteria:

* History of treatment with systemic corticosteroids or hospitalization for a COPD exacerbation in the 4-wk period prior to enrolment.
* Diagnosis of depression or current treatment with antidepressants.
* History of serious psychiatric disorder.
* Myocardial infarction within the last 3 months
* Unstable angina
* Severe cardiac arrhythmia
* Use of any form of smokeless tobacco or nicotine substitution or having followed any cessation program in the past 3 months
* Alcohol or other drug addiction
* Pregnant or lactating women

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Continuous abstinence from week 10 to week 30: This will be defined as self-reported non-smoking combined with an expired CO level ≤ 5 ppm from week 10 through week 30. | week 10 to week 30

SECONDARY OUTCOMES:
Continuous abstinence from week 10 to week 18: This will be defined as self-reported non-smoking combined with an expired CO level ≤ 5 ppm from week 10 through week 18. | week 10 to week 18
Point-prevalence after 3 months and 6 months: This will be defined as abstinence at these time points verified by an exhaled CO level ≤ 5 ppm. | 3 month and 6 month
Motivation to quit: This will be assessed from baseline through quit day. An improvement in motivation in the pre-quitting phase will be defined as an increase in the VAS value from ≤ 3 points at baseline to ≥ 5 points thereafter. | from baseline to week 6
Number of subjects quitting smoking before week 6: The number of subjects quitting smoking at week 4 will be computed for the two groups. | week 4
Differential dropout rate: In order to assess motivational bias this will be calculated at baseline | at baseline
Cigarettes/day: The number of cigarettes smoked per day will be assessed for all participants at all visits. | week 30
Reported smoking reduction: CO level . | from baseline until week 30
  smoking reduction will be defined by decrease in expired CO levels
Decline in pulmonary function: The rate of decline of spirometric parameters will be calculated as the difference between the baseline value and the value observed at end-study. | baseline and week 30
Adverse events: All subjects will be asked about adverse events at each visit by an open-ended question. | week 30
Reported smoking reduction: number of cigarettes. | from baseline until week 30
  smoking reduction will be defined by the reported decrease of number of cigarettes .

CONTACTS AND LOCATIONS:
Overall Officials: Abraham BOHADANA, MD, Principal Investigator — Shaare Zedek Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bohadana A, Rokach A, Wild P, Peker B, Dror YF, Babai P, Arish N, Izbicki G. Varenicline for Gradual Versus Abrupt Smoking Cessation in Poorly Motivated Smokers With COPD: A Prematurely Terminated Randomized Controlled Trial. Chronic Obstr Pulm Dis. 2022 Oct 26;9(4):486-499. doi: 10.15326/jcopdf.2022.0305. PMID 35877930